CLINICAL TRIAL: NCT01821703
Title: A Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LY3045697 After Multiple Oral Dosing in Healthy Subjects
Brief Title: A Study of LY3045697 After Multiple Oral Dosing in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 15051; I6S-MC-ASEB (Other: Eli Lilly and Company); 2013-000475-32 (EudraCT Number)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3045697 (Experimental): Escalating dose (0.1 milligrams [mg] up to 100 mg) of LY3045697 administered once daily, orally, for 8 days in 2 of 3 dosing periods
  Interventions: Drug: LY3045697
- Spironolactone (Active Comparator): 25 mg spironolactone administered once daily, orally, for 8 days in up to 1 of 3 dosing periods
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Placebo matching LY3045697 administered once daily, orally for 8 days in up to 1 of 3 dosing periods
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3045697 — Administered as oral solution
  Arms: LY3045697
Drug: Placebo — Administered as oral solution
  Arms: Placebo
Drug: Spironolactone — Administered as capsule
  Arms: Spironolactone
Drug: Placebo — Administered as capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of LY3045697 after multiple doses and to determine how long LY3045697 remains in the body. Each participant is expected to complete 3 dosing periods. At least 7 days will pass between dosing periods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of non-child bearing potential as determined by medical history and physical examination
* Male participants must agree to use a medically accepted method of contraception with all sexual partners during the study and for 90 days after the end of the final dosing
* Female participants must be postmenopausal or surgically sterile
* Postmenopausal female participants must be between the ages of 45 and 65 years inclusive, and must be 12 months without a menstrual period, or 6-12 months without a menstrual period and Follicle-Stimulating Hormone (FSH) greater than (>)40 International Units per Liter (IU/L)
* Male participants and surgically sterile females are between the ages of 18 and 65 years inclusive
* Have a Body Mass Index (BMI) between 18.0 and 32.5 kilograms per square meter (kg/m2), inclusive, at screening
* Have clinical laboratory test results within normal reference range for the population or investigator site or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow blood sampling
* Are non-smokers or a smoker of 5 or less cigarettes/cigars/pipes per day as determined by history
* Have the ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "power drinks"), poppy seed and tobacco products from 48 hours prior to entry in the clinical research facility until discharge

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 60 days prior to drug administration inclusive from, a clinical trial involving an investigational drug that has not received regulatory approval for any indication
* Have previously completed or withdrawn from this study or any other study investigating this study drug
* Have a history or presence of medical illness including but not limited to any cardiovascular, renal, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, or any clinically significant laboratory abnormality, that in the judgment of the investigator, indicates a medical problem that would preclude study participation
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study, such as a prolonged PR or QRS interval. In addition, participants with the following findings will be excluded:

  * Confirmed corrected QT (QTcF) interval >450 millisecond (msec) for men and >470 msec for women; additional ECGs may be performed if required
  * Complete bundle branch blocks and other conduction abnormalities other than mild first degree atrio-ventricular block
  * Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular ectopic beats
  * History of unexplained syncope
  * Family history of unexplained sudden death or sudden death due to long QT syndrome
  * T-wave configurations are not of sufficient quality for assessing QT interval, as determined by the investigator
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody, or hepatitis B and/or positive hepatitis B surface antigen (HBsAg)
* Intend to use over-the-counter or prescription medication within 5 days prior to dosing, other than daily multi-vitamin therapy, stable thyroid hormone replacement or medication assessed as acceptable by the investigator and not interfering with the integrity of the study data collection. Medications for benign indications in healthy participants may be continued, with the exception of drugs that may alter adrenal function, blood pressure or potassium, such as the use of excessive non-steroidal anti-inflammatory drugs (NSAIDs), glucocorticoids, diuretics, antihypertensive drugs, beta-agonists, and nasal decongestants
* Have donated blood of more than 500 milliliters (mL) within 60 days prior to dosing. Donation of more than 1.5 liters of blood (for men) / more than 1.0 liters of blood (for women) in the 10 months preceding the start of this study (this is the first administration of study drug)
* Have an average weekly alcohol intake that exceeds 21 units per week or participants unwilling to stop alcohol within 48 hours of entry into study until discharge each period [1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Have an abnormal blood pressure (supine) defined as diastolic blood pressure (DBP) >95 or less than (<) 50 millimeter of mercury (mmHg) and/or systolic blood pressure (SBP) >150 or <90 mmHg confirmed by at least 1 repeat measurement
* Regularly use known drugs of abuse or show positive findings for such use on urinary drug screening
* Use of natural licorice (glycyrrhizinic acid) within 5 days of enrollment or use during the study
* Are unwilling to abstain from using grapefruit-containing products and salt-substitutes containing potassium for the duration of the study
* Have known sensitivity or are unable to tolerate spironolactone
* Have serum potassium >upper limit of normal (result from suspected hemolyzed sample may be repeated)
* Have serum sodium <lower limit of normal per lab reference range
* Have serum creatinine >124 micromole/liter (μmol/L) (male); >106 μmol/L (female)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Clinically Significant Adverse Events (AEs) or Any Serious AEs | Baseline to 10 days post last dose (Estimated up to 8 weeks)

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Serum Concentration (Cmax) of LY3045697 | Predose to 24 hours after dosing on Day 8 of each dosing period
Pharmacokinetics: Area Under the Serum Concentration-Time Curve (AUC) from Zero to Infinity (AUC 0-∞) of LY3045697 | Predose to 24 hours after dosing on Day 8 of each dosing period

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zuidlaren, Netherlands